CLINICAL TRIAL: NCT02147691
Title: Finacea 15% and Brimonidine 0.33% Gel in the Treatment of Rosacea - A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Principal Investigator, Leon Kircik, M.D., Medical Director, Derm Research, PLLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIN1302
Record Dates: First submitted 2014-05-16; First posted 2014-05-28 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-08

CONDITIONS: Acne Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azelaic acid 15%, Brimonidine 0.33 % Gel (Experimental): Azelaic acid 15% to the face each AM followed 30 minutes later by Brimonidine 0.33%
  Azelaic acid 15% to the face each PM
  Interventions: Drug: Azelaic acid 15%; Drug: Brimonidine 0.33%
- Brimonidine 0.33% Gel (Active Comparator): Brimonidine 0.33% Gel
  Interventions: Drug: Brimonidine 0.33%

INTERVENTIONS:
Drug: Azelaic acid 15% — Applied to the face each AM and PM
  Other Names: Finacea
  Arms: Azelaic acid 15%, Brimonidine 0.33 % Gel
Drug: Brimonidine 0.33% — Applied to the face each AM 30 minutes after the application of Azelaic acid 15%
  Other Names: Miravaso

SUMMARY:
The pilot study will investigate whether combination treatment of Finacea 15% Gel and Brimonidine 0.33% Gel could be more effective than Brimonidine 0.33% Gel monotherapy in treating both the papules/pustules and erythema associated with rosacea.

DETAILED DESCRIPTION:
Acne rosacea is a chronic inflammatory disease with different components including inflammatory lesions (papules/pustules), erythema and telangiectasia. Brimonidine 0.33% Gel primarily affects the erythematous components of rosacea. As such, combination treatment with a standard rosacea treatment, such as Finacea 15% Gel, may provide additional relief for the inflammatory component of rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 years of age and older
* Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline
* Female subjects of childbearing potential must practice a reliable method of contraception throughout the study
* Moderate or severe rosacea with an Investigator Global Assessment (IGA) score of 3 or 4
* Able to understand and comply with the requirements of the study and sign Informed Consent/Health Insurance Portability and Accountability Authorization forms

Exclusion Criteria:

* Female subjects who are pregnant, breast feeding or who are of childbearing potential and not practicing a reliable method of birthcontrol
* History of hypersensitivity or idiosyncratic reaction to any component of the test medications
* Subjects who have not completed the proper wash-out periods for prohibited medications and/or procedures
* Medical condition that contraindicates the subject's participation in the study
* Alcohol or drug abuse is evident within the past 5 years
* History of poor cooperation, non-compliance with medical treatment, unreliability
* Participation in an investigational drug study within 30 days of the Baseline visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H. Kircik, M.D., Principal Investigator — DermResearch, PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single site recruitment, private medical clinic.. Subjects 18 to 85 years of age with moderate to severe rosacea.Recruitment began May 2014 and ended November 2014.
Pre-assignment Details: Subjects could be excluded if less than 18 years of age, who does not have moderate to severe rosacea as determined by the Investigator Global Assessment (IGA), who has not completed the specified washout for medications as outlined in the protocol or who has been in another investigational study within 30 days of the Baseline visit.
Groups:
- Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 0.33 % Gel: Finacea 15% Gel (azelaic acid 15%) followed 30 minutes later with application of Brimonidine 0.33% Gel each morning to the face
  Finacea 15 % Gel (azelaic acid 15%) each evening to the face
  Azelaic acid 15%
  Brimonidine 0.33%
- Brimonidine 0.33% Gel: Brimonidine 0.33% Gel applied to the face each morning
  Brimonidine 0.33%
Period: Overall Study
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 0.33 % Gel | Brimonidine 0.33% Gel
Started | 10 | 12
Completed | 6 | 11
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: subjects between 18 years and 85 years of age with moderate to severe rosacea
Groups:
- Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel: Finacea 15% Gel (azelaic acid 15%) followed 30 minutes later with application of Brimonidine 0.33% Gel each morning to the face
  Finacea 15 % Gel (azelaic acid 15%) each evening to the face
  Azelaic acid 15%
  Brimonidine 0.33%
- Total: Total of all reporting groups
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 11 | 17
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (IGA) at Baseline
Description: Assessment of rosacea on a scale of 0-4, 0 = clear, 1= almost clear, 2= mild, 3= moderate and 4 = severe
Time Frame: Baseline
Population: Only participants who were not lost to follow up or did not withdraw consent were included in the final analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Brimonidine 0.33% Gel: Brimonidine 0.33% Gel applied to the face each morning
  Brimonidone 0.33%
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 3 (0) | 3.1 (0.3)

2. Secondary Outcome: Lesion Counts
Description: The number of inflammatory lesions (papules/pustules) will be counted using the whole face from the hairline edge to the mandibular line
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
lesions | 3.3 (1.6) | 4.5 (2.8)

3. Secondary Outcome: Clinician's Erythema Assessment
Description: Erythema will be graded on a scale of 0-4., 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 very severe. If erythema is much worse on one or several parts of the face, the grade for the worst area will be captured.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 2.3 (0.5) | 2.1 (0.3)

4. Secondary Outcome: Erythema Visual Analog Scale (VAS) Assessment (Subject)
Description: Subjects will self assess the level of erythema over the previous 24 period using a scale of None (0) through 10 (Unbearable)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 5.5 (2.5) | 5.6 (1.8)

5. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: The DLQI is a self-administered questionnaire consisting of 10 questions that measure how much the individual's skin problem has affected their life in the past week. Score ranges 0 through 30, 0 being none and 30 worst possible.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 2.6 (3.7) | 2.9 (1.9)

6. Primary Outcome: IGA
Description: Assessment of rosacea on a scale of 0-4, 0 = clear, 1= almost clear, 2= mild, 3= moderate and 4 = severe
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.8 (0.9) | 1.8 (0.8)

7. Primary Outcome: IGA
Description: Assessment of rosacea on a scale of 0-4, 0 = clear, 1= almost clear, 2= mild, 3= moderate and 4 = severe
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.6 (1.2) | 1.8 (0.9)

8. Primary Outcome: IGA
Description: Assessment of rosacea on a scale of 0-4, 0 = clear, 1= almost clear, 2= mild, 3= moderate and 4 = severe
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.3 (1.1) | 1.4 (0.9)

9. Secondary Outcome: Lesion Count
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
lesions | 1.1 (1.2) | 2.1 (2.9)

10. Secondary Outcome: Lesion Counts
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
lesions | 1.0 (1.4) | 1.7 (2.1)

11. Secondary Outcome: Lesion Counts
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
lesions | 0.7 (1.3) | 1.2 (1.3)

12. Secondary Outcome: Erythema
Description: Erythema as measured by the clinician on a scale of 0-4, 0 = no erythema, 1 = slight pinkness, 2 = moderate, definite redness, easily recognized, 3 = severe, marked erythema and 4 = very severe, fiery red
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.6 (0.7) | 1.3 (0.7)

13. Secondary Outcome: Erythema
Description: as for outcome 12
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.3 (0.8) | 1.4 (0.7)

14. Secondary Outcome: Erythema
Description: as for outcome 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.3 (0.7) | 1.2 (0.8)

15. Secondary Outcome: Visual Analog Scale (VAS)
Description: participant measures erythema on a scale of 0 mm to 10 mm with 0 = to none and 10 = unbearable
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 4.5 (2.4) | 5.2 (2.1)

16. Secondary Outcome: VAS
Description: participant measures erythema on a scale of 0 mm to 10 mm with 0 = to none and 10 = unbearable
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 4.4 (3.0) | 4.5 (2.1)

17. Secondary Outcome: VAS
Description: participant measures erythema on a scale of 0 mm to 10 mm with 0 = to none and 10 = unbearable
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 3.8 (2.3) | 4.0 (2.1)

18. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: Total scores range from 0 ( no impact on life over the last week) to 30 (maximum impact on life over the last week)
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.8 (1.5) | 2.6 (2.0)

19. Secondary Outcome: DLQI
Description: Total scores range from 0 ( no impact on life over the last week) to 30 (maximum impact on life over the last week)
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.3 (1.2) | 2.6 (2.6)

20. Secondary Outcome: DLQI
Description: Total scores range from 0 ( no impact on life over the last week) to 30 (maximum impact on life over the last week)
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Number analyzed (Participants) | 6 | 11
units on a scale | 1.2 (1.2) | 2.8 (2.8)

ADVERSE EVENTS:
Arm/Group | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel | Brimonidine 0.33% Gel
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 3/10 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finacea 15% Gel (Azelaic Acid 15%), Brimonidine 15 % Gel (N=10) | Brimonidine 0.33% Gel (N=12)
pulled muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — right hip
Broken toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Left fourth toe
worsening erythema on face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — treatment area
worsening facial lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — treatment area
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
common cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
herpes simplex (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Adjacent to treatment area
burning at application site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Pilot study. Small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes